CLINICAL TRIAL: NCT00169208
Title: An Open Label, Multicenter, Non Randomized Phase II Study to Evaluate Anti-tumor Activity and Safety of a Combination of Fludarabine, Mitoxantrone and Rituximab in Relapsed or Primary Failing Advanced Follicular Non-Hodgkin's Lymphoma.
Brief Title: Fludarabine, Mitoxantrone and Rituximab in Relapsed or Primary Failing Advanced Follicular Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lymphoma Study Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RFM Follicular lymphoma study
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Follicular Lymphoma
Keywords: relapsed/refractory.; lymphoma, follicular; rituximab; chemotherapy
MeSH Terms: conditions — Lymphoma, Follicular; Recurrence | interventions — Rituximab; fludarabine; Mitoxantrone

ARMS (1):
- Experimental (Experimental): 4 cycles of rituximab + fludarabine + mitoxantrone
  Interventions: Drug: rituximab; Drug: fludarabine; Drug: mitoxantrone

INTERVENTIONS:
Drug: rituximab — 375 mg/m² IV, D1 each cycle during 4 cycles
Drug: fludarabine — 40 mg/m²/day IV , D1 each cycle during 4 cycles
Drug: mitoxantrone — 10 mg/m² IV, D2-3-4 each cycle during 4 cycles

SUMMARY:
This study is a multicentric trial evaluating the efficacy of the RFM regimen in patients aged 18 to 75 years with relapsed/refractory follicular non-Hodgkin's lymphoma (NHL).

DETAILED DESCRIPTION:
Follicular non Hodgkin's lymphoma's (FL), as defined by the Revised European American Lymphoma Classification (REAL) Classification, are usually characterized by a slowly progressive clinical course, a transient control by standard chemotherapeutic regimen and a pattern of repeated relapses until ultimately progressive and fatal disease.

Standard first line treatment for advanced FL consists of alkylating-based (CVP) or anthracycline containing regimen in association to interferon alpha (CHVP+IFN) chemotherapy. Others approaches have been developed mostly as secondary therapy including purine analogs alone or in combination with alkylators or mitoxantrone, high dose therapy with autologous peripheral stem cell transplantation and, more recently, treatment with the unconjugated chimeric anti-CD20 antibody (rituximab) to target the CD20 antigen highly expressed on follicular lymphoma cells. None of these strategies does appear to give a definitive survival advantage. Thus, in patients with FL, the design of novel combination programs is a major challenge.

Combination of fludarabine and mitoxantrone in low grade, predominantly Follicular NHL: results of phase II studies in relapsed or refractory patients Fludarabine is expected to potentiate other agents through inhibition of DNA polymerase alpha and DNA ligase and its consequent interference with the DNA repair process. The addition of mitoxantrone increases the cytotoxic effect of fludarabine in vitro. McLaughlin et al developed a combination of fludarabine, mitoxantrone and dexamethasone (FND), which was very effective in 51 patients with recurrent low-grade lymphoma (including 65% FL), with an overall response rate of 94% (47% complete response (CR) rate. The median duration of response in this phase II study was 21 months for CR patients but only 9 months for partial responders (PR) patients. The median survival and failure-free survival times from the time of entry onto the FND study were 34 and 14 months, respectively. Most major responses were evident after two to four courses of chemotherapy. The need for continuation of therapy beyond attainment of remission is suggested by early relapses among patients who had early discontinuation of therapy. The predominant toxic effects were myelosuppression and infections: neutropenia < 500/µl in 20 % of courses, thrombopenia < 50000/µl in 8 % of courses and infections in 12 % of courses. Non-hematological toxicity was modest.

FND appears to be comparable to, and less toxic than the combination of etoposide, methylprednisolone, cytarabine, and cisplatin (ESHAP), one of the most effective regimens available for patients with relapsed indolent lymphoma. Others studies have confirmed the significant efficacy and moderate toxicity profile of this combination as salvage therapy in low grade, predominantly follicular lymphoma.

Moreover, the omission of corticosteroids reduces the risk of opportunistic infections, while the activity of the combination against indolent lymphoma is maintained.

Preliminary data from rituximab studies alone or in combination with chemotherapy in relapsed or refractory low grade NHL In vitro, rituximab mediates complement dependent cytotoxicity (CDC), antibody dependent cellular cytotoxicity (ADCC) and apoptosis. However, the mechanism of in vivo anti-lymphoma effect remains largely unknown. Rituximab received approval for recurrent follicular lymphoma based on response rates of about 50% including 6% complete responses and duration of responses, which compare favorably to that of all other single agents including fludarabine and 2-CdA (15-19). Median time to progression for responders is around 13 months. Toxicity of rituximab is low and easily manageable. An 8 doses schedule did not show to confer a significant advantage in term of response rate and duration of response over the four doses schedule.

Rituximab has been shown to sensitize drug-resistant lymphoma cell lines to killing by cytotoxic drugs including fludarabine.

Thus, we may hypothesize that the combination of rituximab, fludarabine and mitoxantrone might lead to synergistic / additive induction of apoptosis through different pathways in lymphoma B-cells which maintain an indolent growth pattern.

This approach may provide a means to achieve longer progression free survival in relapsed or refractory patients with FL.

We opted for a four induction cycles of rituximab, fludarabine and mitoxantrone since:

1. Four cycles of a combination of fludarabine and mitoxantrone are generally sufficient to assess response,
2. the 4 doses schedule of rituximab which has been the most studied is efficient 3) The omission of dexamethasone does not appear to impair ORR and Duration Response (DR) of a combination of fludarabine and novantrone . Recycling will start on day 28.

Subsequently responding patients according the International criteria Working group will have 2 more cycle of a combination of fludarabine and mitoxantrone but no rituximab.

ELIGIBILITY:
Inclusion Criteria:

* 18 years < age < 75 years
* Pathologically confirmed low grade, follicular, B cell lymphoma (WHO Classification Follicular grades 1 and 2
* Failed at least first line chemotherapy with any standard anthracycline containing regimen (see appendix C for definition of treatment failure)
* Frozen biopsy material obtained at relapse or disease progression should be available for central pathology review and molecular biology studies
* The lymphoma must be CD20 positive (on the biopsy material obtained at relapse or disease progression)
* At least one measurable lesion one nodal or extranodal lesion
* WHO performance status grade 0 or 1
* Bulky disease at study entry according to the Groupe d'Etude des Lymphomes Folliculaires (GELF) criteria: Nodal or extranodal single mass > 7cm in its greatest diameter; systemic B-symptoms; increased lactate dehydrogenase (LDH) and beta 2 macroglobulinemia (> 3mg/L); involvement of at least 3 nodal sites, each with a diameter of greater than 3 cm; splenic enlargement with margin below the umbilical line or cranio caudal diameter of greater than 20 cm; compression syndrome (ureteral, orbital, gastrointestinal), or pleural or peritoneal serous effusion.
* Patient information and written informed consent

Exclusion Criteria:

* Evidence of histological transformation to diffuse large B-cell lymphoma
* > 2 prior treatment regimen
* Chemotherapy, or other experimental anticancer treatment during the 4 weeks before inclusion
* Any radiation therapy to the index lesion(s) during the 4 weeks before inclusion
* Autologous stem cell transplant during the 3 months before inclusion
* Prior treatment including fludarabine and / or mitoxantrone and / or rituximab or contra-indication to one of these products
* Unless exempted by the Responsible Investigator, as lymphoma related: serum creatinine >2 x Institutional Upper Limit of Normal (IULN), total bilirubin >2 x IULN or aspartate aminotransferase (AST) >2 x IULN, alkaline phosphatase >2 x IULN
* Low bone marrow function: absolute neutrophil count < 1500/mm3 and platelet < 100 x 109/L at study entry (unless bone marrow infiltration)
* Clinically significant cardiac disease, as defined by history of symptomatic ventricular arrhythmias, congestive heart failure or myocardial infarction within 12 months of study entry
* Evidence of symptomatic central nervous system disease
* Known positivity for HIV, hepatitis Bs antigen or hepatitis C
* Pregnant or lactating women. Women of childbearing potential, and all men, unwilling to take appropriate contraceptive measures during and for at least 6 months after cessation of therapy
* Patients considered for an autologous or allogenic stem transplant at time of primary treatment failure or relapse according to the rules of the respective centers
* Any uncontrolled serious non malignant condition or infection which would likely compromise the study objectives
* Previous evolutive malignancy within 5 years of study entry, with the exception of non-melanoma skin tumors or stage 0 (in situ) cervical carcinoma
* Major surgery within 4 weeks prior to enrollment, unless patient has recovered from all treatment related toxicity
* Patient under tutelage.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2001-04 (Actual); Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
to evaluate progression free survival after a combination of rituximab, fludarabine and mitoxantrone (RFM) in patients with relapsed or primary failing advanced follicular non-Hodgkin's lymphoma. | 2 years

SECONDARY OUTCOMES:
overall response rate (ORR) | 5 years
complete response (CR) | 5 years
to evaluate overall survival (OS) | 5 years
duration of response | 5 years
number of Serious Adverse Event (SAE) | 5 years
to monitor minimal residual disease using the molecular biological marker bcl2 in peripheral blood and bone marrow | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Franck Morschhauser, MD, Principal Investigator — Lymphoma Study Association; Charles FOUSSARD, MD, Study Chair — French Innovative Leukemia Organisation
Locations (16):
- France (16):
  - Service de médecine D - Maladies du Sang CHU Angers, Angers
  - Service d'Hématologie Hôpital Jean Minjoz, Besançon
  - Hôpital Henri Mondor, Créteil
  - Hôpital A. Michallon BP 217X, Grenoble
  - Service Oncologie - Centre Victor Hugo, Le Mans
  - Service d'hématologie clinique - Centre Hospitalier du Dr Schaffner, Lens
  - Hôpital Claude Huriez - Sce des Maladies du Sang - Place Verdun, Lille
  - Centre Hospitalier Lyon-sud, Lyon
  - Centre régional de lutte contre le cancer Léon Bérard, Lyon
  - Service d'hématologie Institut Paoli Calmette, Marseille
  - Service d'hématologie - Hôpital Necker, Paris
  - Service d'Hématologie Hôpital St Louis, Paris
  - Service d'hématologie clinique - Hôpital de Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen
  - Service Oncologie CHU Bretonneau, Tours
  - Service d'hématologie Institut Gustave Roussy, Villejuif

REFERENCES:
- [Background] Horning SJ. Natural history of and therapy for the indolent non-Hodgkin's lymphomas. Semin Oncol. 1993 Oct;20(5 Suppl 5):75-88. No abstract available. PMID 8211209
- [Background] McLaughlin P, Hagemeister FB, Romaguera JE, Sarris AH, Pate O, Younes A, Swan F, Keating M, Cabanillas F. Fludarabine, mitoxantrone, and dexamethasone: an effective new regimen for indolent lymphoma. J Clin Oncol. 1996 Apr;14(4):1262-8. doi: 10.1200/JCO.1996.14.4.1262. PMID 8648382
- [Background] Maloney DG, Grillo-Lopez AJ, White CA, Bodkin D, Schilder RJ, Neidhart JA, Janakiraman N, Foon KA, Liles TM, Dallaire BK, Wey K, Royston I, Davis T, Levy R. IDEC-C2B8 (Rituximab) anti-CD20 monoclonal antibody therapy in patients with relapsed low-grade non-Hodgkin's lymphoma. Blood. 1997 Sep 15;90(6):2188-95. PMID 9310469
- [Result] McLaughlin P, Grillo-Lopez AJ, Maloney DG, Link BK, Levy R, Czuczman MS, Cabanillas F, Dallaire BK, White CA: Efficacy controls and long-term follow-up of patients treated with rituximab for relapsed or refractory, low-grade or follicular NHL. Blood 92:414a, 1998
- See also: Official site of the Groupe d'Etudes des Lymphomes de l'Adulte (In french) — http://www.gela.org